CLINICAL TRIAL: NCT03690713
Title: International Patient-level Pooled Analysis of Comprehensive Physiologic Assessment: Collaborating Project of Korea, Japan, and Spain
Brief Title: International Collaboration of Comprehensive Physiologic Assessment
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Samsung Medical Center (Other); Tsuchiura Kyodo General Hospital (Other); Hospital San Carlos, Madrid (Other); Imperial College Healthcare NHS Trust (Other); Tokyo Medical and Dental University (Other); Sungkyunkwan University (Other); Inje University (Other); Keimyung University Dongsan Medical Center (Other); Ulsan University Hospital (Other)
Responsible Party: Principal Investigator, Bon-Kwon Koo, Professor, Seoul National University Hospital
Other Study IDs: NCT186918690001
Record Dates: First submitted 2018-09-26; First posted 2018-10-01 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Stable Angina; Unstable Angina; Non-ST Elevation Myocardial Infarction; ST-segment Elevation Myocardial Infarction
Keywords: fractional flow reserve; myocardial ischemia; coronary artery disease; coronary flow reserve; index of microcirculatory resistance; prognosis; percutaneous coronary intervention
MeSH Terms: conditions — Angina, Stable; Angina, Unstable; Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction; Myocardial Ischemia; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient and Vessels underwent physiologic evaluation: The total 1397 patients (1694 vessels) which evaluated using pressure-temperature sensor wire and measured FFR, CFR, and IMR.
  Interventions: Diagnostic Test: Fractional flow reserve, coronary flow reserve, and index of microcirculatory resistance

INTERVENTIONS:
Diagnostic Test: Fractional flow reserve, coronary flow reserve, and index of microcirculatory resistance — The pressure sensor was positioned at the distal segment of a target vessel, and intracoronary nitrate was administered before each physiologic measurement. To derive resting mean transit time (Tmn), a thermodilution curve was obtained by using 3 injections (3-4 mL each) of room-temperature saline. Hyperemic proximal aortic pressure (Pa), distal arterial pressure (Pd), and hyperemic Tmn were measured during sustained hyperemia. CFR was calculated as resting Tmn/hyperemic Tmn. FFR was calculated as the lowest average of 3 consecutive beats during hyperemia. The uncorrected IMR was calculated by Pd × Tmn during hyperaemia. All IMR values were corrected by Yong's formula (Pa × Tmn × ([1.35 × Pd/Pa] - 0.32).

SUMMARY:
The current study evaluated prognostic implication of comprehensive physiologic assessment using fractional flow reserve, coronary flow reserve (CFR) and index of microcirculatory resistance (IMR).

DETAILED DESCRIPTION:
The patient-level data was gathered from 3 nations (Korea, Japan, Spain). The total 1397 patients (1694 vessels) data was collected from 5 university hospitals in Korea (Seoul National University Hospital, Samsung Medical Centre, Inje University Ilsan Paik Hospital, Keimyung University Dongsan Medical Centre, and Ulsan University Hospital, Korea) and Tsuchiura Kyodo General Hospital, Ibaraki, Japan, and Hospital Clinico San Carlos, Madrid, Spain.

Standardized form of data collection sheet was used and all study adopted standardized definition of patient's baseline characteristics, clinical outcomes, and physiologic data. In case of acute coronary syndrome (unstable angina, non-ST-segment elevation myocardial infarction, and ST-segment elevation myocardial infarction), only non-culprit vessel was included in the data.

Primary outcome is patient- and vessel-oriented composite outcome at 5 years.

ELIGIBILITY:
Inclusion Criteria:

- patients who underwent clinically indicated invasive coronary angiography and measurements of FFR, CFR, and IMR for at least 1 coronary artery

Exclusion Criteria:

* Patients with hemodynamic instability
* left ventricular dysfunction
* culprit vessel of acute coronary syndrome

Age Groups: Child, Adult, Older Adult
Study Population: patients who underwent clinically indicated invasive coronary angiography and measurements of FFR, CFR, and IMR for at least 1 coronary artery
Sampling Method: Non-Probability Sample
Enrollment: 1397 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
Cumulative incidence of a composite of any death, any myocardial infarction, or any ischemia-driven revascularization | 5 year
  Patient-oriented composite outcome
Cumulative incidence of a composite of cardiac death, target-vessel related myocardial infarction, or target-vessel revascularization | 5 year
  Vessel-oriented composite outcome

SECONDARY OUTCOMES:
Cumulative incidence of any death | 5 year
  all-cause mortality
Cumulative incidence of cardiac death | 5 year
  cardiac death
Cumulative incidence of myocardial infarction | 5 year
  MI was defined as elevated cardiac enzyme levels greater than the upper limit of the normal range with either ischemic symptoms or electrocardiography changes indicating ischemia after index procedure. Periprocedural MI was not included as a clinical outcome
Cumulative incidence of ischemia-driven revascularization | 5 year
  Ischemia-driven revascularization was defined as a revascularization procedure with at least one of the following: (1) recurrence of angina; (2) positive non-invasive test; and (3) positive invasive physiologic test

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon Koo, MD, PhD, Study Chair — Seoul National University Hospital; Javier Escaned, MD, PhD, Study Chair — Hospital Clinico San Carlos, Madrid, Spain; Tsunekazu Kakuta, MD, PhD, Study Chair — Tokyo Medical and Dental University, Tokyo, Japan; Joo Myung Lee, MD, MPH, PhD, Study Chair — Samsung Medical Center, Seoul, Korea
Locations (4):
- Tokyo Medical and Dental University, Tokyo, Japan
- South Korea (2):
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Hospital Clinico San Carlos, Madrid, Spain, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Anonymized patient level data will be made available by the corresponding author for reasonable requests. Consent was not obtained for data sharing but the presented data are anonymized and risk of identification is minimal.

REFERENCES:
- [Derived] Shin D, Lee JM, Lee SH, Hwang D, Choi KH, Kim HK, Doh JH, Nam CW, Shin ES, Hoshino M, Murai T, Yonetsu T, Mejia-Renteria H, Kakuta T, Escaned J, Koo BK. Non-randomized comparison between revascularization and deferral for intermediate coronary stenosis with abnormal fractional flow reserve and preserved coronary flow reserve. Sci Rep. 2021 Apr 28;11(1):9126. doi: 10.1038/s41598-021-88732-4. PMID 33911143
- [Derived] Lee JM, Choi KH, Doh JH, Nam CW, Shin ES, Hoshino M, Murai T, Yonetsu T, Mejia-Renteria H, Kakuta T, Escaned J, Koo BK. Long-term Patient Prognostication by Coronary Flow Reserve and Index of Microcirculatory Resistance: International Registry of Comprehensive Physiologic Assessment. Korean Circ J. 2020 Oct;50(10):890-903. doi: 10.4070/kcj.2020.0083. Epub 2020 May 27. PMID 32725991
- [Derived] Hamaya R, Lee JM, Hoshino M, Yonetsu T, Koo BK, Escaned J, Kakuta T; Collaborators. Clinical outcomes of Fractional Flow Reserve-Guided Percutaneous Coronary Intervention By Coronary Flow Capacity Status in Stable Lesions. EuroIntervention. 2021 Jul 20;17(4):e301-e308. doi: 10.4244/EIJ-D-20-00401. PMID 32624458
- [Derived] Hamaya R, Hoshino M, Yonetsu T, Lee JM, Koo BK, Escaned J, Kakuta T. Defining heterogeneity of epicardial functional stenosis with low coronary flow reserve by unsupervised machine learning. Heart Vessels. 2020 Nov;35(11):1527-1536. doi: 10.1007/s00380-020-01640-x. Epub 2020 Jun 6. PMID 32506182
- [Derived] Lee SH, Lee JM, Park J, Choi KH, Hwang D, Doh JH, Nam CW, Shin ES, Hoshino M, Murai T, Yonetsu T, Mejia-Renteria H, Kakuta T, Escaned J; International Collaboration of Comprehensive Physiologic Assessment Investigators. Prognostic Implications of Resistive Reserve Ratio in Patients With Coronary Artery Disease. J Am Heart Assoc. 2020 Apr 21;9(8):e015846. doi: 10.1161/JAHA.119.015846. Epub 2020 Apr 18. PMID 32306809